CLINICAL TRIAL: NCT01402115
Title: Efficacy and Safety Study of Polycan on Bone Metabolism
Brief Title: A 12-week Human Trial to Compare the Efficacy and Safety of Polycan on Bone Metabolism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Glu-POLYCAN-001
Record Dates: First submitted 2011-07-21; First posted 2011-07-26 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Bone Health in Perimenopausal Women
Keywords: Polycan; Bone metabolism; Osteocalcin; Deoxypyridinoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polycan (Experimental): Polycan 150mg for 12 weeks
  Interventions: Dietary Supplement: Polycan
- Placebo (Placebo Comparator): Placebo 15mg for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Polycan — polycan 150 mg/d for 12 weeks
  Arms: Polycan
Dietary Supplement: Placebo — Placebo 150mg/d for 12 weeks
  Arms: Placebo

SUMMARY:
Beta-glucans are polysaccharides consisting of glucose residue jointed by beta linkage. They are found at a high level in the cell wall of fungi, yeast, oat, barley, bacteria, as well as various mushroom. Studies have reported that extract of mushroom (Pleurotus eryngii) can prevent the bone loss caused by estrogen deficiency. Furthermore, polycan (a purified β-glucan from Aureobasidium pullulans) has been reported to exhibit osteoporosis preventing effects. However, no investigation has been conducted on the effect of polycan on bone health in perimenopausal women.

Therefore, in this study, we investigated the effect of polycan on biochemical markers of bone metabolism in Korean perimenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* They were required to have reduced bone density but no evidence of osteoporosis or osteopenia by Dual-emission X-ray absorptiometry (DEXA) scan (T ≥ -1.0 in the lumbar spine).
* Perimenopausal women : aged 40-70

Exclusion Criteria:

* Women with a body mass index (BMI) >30 kg/m2 or who were being treated with estrogens, corticosteroids, or bisphosphonates, or who had significant illness affecting bone metabolism were excluded

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dal-Sik Kim, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Healthcare claims and management; Chonbuk National university, Jeonju, Jeollabuk-do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through local advertising and doctor referrals from hospital outpatients and general practice clinics.
Pre-assignment Details: The criteria were an age from 40 to 70 years, They were required to have reduced bone density but no evidence of osteoporosis or osteopenia by Dual-emission X-ray absorptiometry (DEXA) scan (T ≥ -1.0 in the lumbar spine).
Period: Overall Study
Arm/Group | Polycan | Placebo
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polycan | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52.8 (6.3) | 52.9 (5.8) | 52.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Changes in DPD(Deoxypyridinoline)
Description: DPD(Deoxypyridinoline) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: nanoMolar DPD per milliMolar creatine
Arm/Group | Polycan | Placebo
Number analyzed (Participants) | 29 | 29
nanoMolar DPD per milliMolar creatine
  Pre | 7.1 (2.2) | 6.4 (1.7)
  Post | 6.2 (2.1) | 5.6 (1.5)

2. Primary Outcome: Changes in OSC(Osteocalcin)
Description: OSC(Osteocalcin) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Polycan | Placebo
Number analyzed (Participants) | 29 | 29
ng/mL
  Pre | 16.1 (6.8) | 14.2 (5.2)
  Post | 19.8 (7.7) | 17.0 (6.8)

3. Secondary Outcome: Changes in CTx(Collagen Type 1 Cross-linked C-telopeptide)
Description: CTx(collagen type 1 cross-linked C-telopeptide) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Polycan | Placebo
Number analyzed (Participants) | 29 | 29
µg/L
  Pre | 344 (183) | 314 (217)
  Post | 341 (171) | 301 (157)

4. Secondary Outcome: Changes in bALP(Bone-specific Alkaline Phosphatase)
Description: bALP(bone-specific alkaline phosphatase) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Polycan | Placebo
Number analyzed (Participants) | 29 | 29
U/L
  Pre | 31.8 (11.3) | 28.6 (9.7)
  Post | 31.8 (11.7) | 29.8 (9.5)

5. Secondary Outcome: Changes in PTH(Parathyroid Hormone)
Description: PTH(parathyroid hormone) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Polycan | Placebo
Number analyzed (Participants) | 29 | 29
pg/mL
  Pre | 32.8 (10.4) | 31.1 (8.7)
  Post | 35.0 (9.3) | 33.6 (7.5)

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Polycan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No